CLINICAL TRIAL: NCT06804109
Title: Vaping and Vagal Neuromodulation of Cognition
Brief Title: Non-invasive Vagus Nerve Stimulation (nVNS) and Cognition in Young Adult Vapers - A Pilot Study
Acronym: nVNS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB31783
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Vaping
Keywords: vaping; attention; non-invasive vagus nerve stimulation
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Active Stimulation (Experimental): Participants in the active arm will receive a 2-min transcutaneous vagus nerve stimulation using a portable hand-held digital wellness Truvaga Plus device by placing it on the anterolateral cervical area of the neck.
  Interventions: Device: Active nVNS
- Control Stimulation (Experimental): Participants in the control arm will receive a 2-min transcutaneous stimulation using a portable hand-held digital wellness Truvaga Plus device by placing it on the posterolateral part of the neck (near the overlapping area between the trapezeus muscle and the shoulder).
  Interventions: Device: Control nVNS

INTERVENTIONS:
Device: Active nVNS — 2-min transcutaneous nVNS stimulation using portable Truvaga Plus Device (electroCore Inc., Rockaway, NJ).
  Arms: Active Stimulation
Device: Control nVNS — 2-min control stimulation using portable Truvaga Plus Device (electroCore Inc., Rockaway, NJ).
  Arms: Control Stimulation

SUMMARY:
The purpose of this study is to assess the effects of non-invasive vagus nerve stimulation (nNVS) on cognitive functioning in the users of e-cigarettes or vaping products. The investigators will use a digital wellness companion product (TRUVAGA™ device) that provides mild transcutaneous nVNS. The participants will be randomized to receive either a 2-min nNVS stimulation or control stimulation in the neck region followed by completion of three cognitive tests of attention and executive function.

DETAILED DESCRIPTION:
Electronic cigarettes, also referred to as e-cigarettes or vapes were initially developed as a smoking cessation tool and considered less harmful, but the presence of nicotine in the vapes make them highly addictive. The use of E-cigarettes has dramatically increased among the youth and young adults in the last decade. While the risks associated with traditional, combustible cigarette smoking are "well-established," vaping also exposes individuals to nicotine which is highly addictive and it can have long-term detrimental effects on the brain. Impairments in cognitive processes including attention and executive functions are suggested to contribute to the development and maintenance of sustained nicotine use in addicts and improving these processes may have some benefits. One of the ascending neuromodulatory input system, the cholinergic system, is implicated in the regulation of attention and higher-order cognitive processes. The stimulation of peripheral vagus nerve is known to activate ascending neuromodulators in the brain including the cholinergic system. This pilot project will use a single blind between-subjects randomized design to investigate the effects of non-invasive vagus nerve stimulation (nNVS) on attentional capacities in e-cigarette users. The study will involve administration of self-report surveys regarding vaping dependence and craving, measures of attention, impulsivity, anxiety and negative emotional states, and two quick behavioral tests (reaction time and lexical retrieval) to assess baseline measures of processing speed and executive function. For baseline processing speed assessment, the participants will complete a quick (3-5 min) simple and choice Reaction Time task on a computer prior to the intervention. The lexical retrieval efficiency will be assessed by 1-min Verbal Fluency Test prior to the intervention. Following this, the participants will be randomized to receive either a 2-min nNVS stimulation or control stimulation in the neck region using a portable TruvagaTM Plus device (electroCore). This digital device is a general health and wellness (Digital Health) product and is not intended to diagnose, cure, mitigate, treat, or prevent any disease. The subjects will complete three neuropsychological tests of attention and executive function (Attention Network Test, Symbol Digit Modalities Test, and Verbal Fluency Test) immediately after the intervention. The 1-min Verbal Fluency Test will be completed by the participants both before (pre-test) and after (post-test) the intervention. The specific goals of the study are: 1) To test the hypothesis that e-cigarette users given acute transcutaneous nNVS will perform better on tasks of attention as compared to e-cigarette users given control stimulation. 2): To test the hypothesis that cognitive benefits of nNVS in e-cigarette users will be associated with the degree of nicotine dependence and the magnitude of negative affective states.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young adults
* Age range 18-25 years
* Current or prior users of e-cigarettes

Exclusion Criteria:

Participants will be excluded from the study if they:

* Have any rash, infection, swelling, cut, soreness, drug patch, surgical scar on the neck area
* Have any implantable medical device in their body such as a pacemaker, hearing aid implant, or any other metallic/electronic device
* Have any hearing or vision problems that are not corrected
* Are pregnant or breastfeeding
* Have any learning disabilities
* Have a medical history of any of the following condition
* Meningitis
* Traumatic brain injury
* Seizure
* Syncope
* Schizophrenia
* Schizoaffective disorder
* Bulimia (eating disorder)
* Other serious neurological illness
* Have a medical history of any of the following cardiac disorder

  * Carotid atherosclerosis or carotid artery disease
  * Cervical vagotomy
  * First degree atrioventricular block or prolonged QT interval
* Are taking any medications for to treat hypertension, arrhythmias, or are on calcium channel blockers

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2027-02-09 (Estimated); Study Completion 2028-02-09 (Estimated)

PRIMARY OUTCOMES:
Efficiency of Attentional Networks using the Attention Network task (ANT) | Immediately after intervention
  The Attentional Network Task (ANT) measures alerting, orienting, and executive attention that combines spatial cues with different flanker conditions. The efficiency of these three attentional networks is assessed by averaging reaction times and accuracy.
Attention and Processing Speed using the Symbol Digit Modalities Test (SDMT) | Immediately after intervention
  The Symbol Digit Modalities Test (SDMT) is a sensitive and reliable neuropsychological test for the evaluation of speed of information processing, scanning and tracking aspects of attention, and working memory. SDMT is a simple substitution task that uses a reference key for the participants to pair specific numbers with given geometric figures. The test score is calculated based on the number of correct responses in 90 seconds.
Lexical Retrieval using the Verbal Fluency Task | Before and immediately after the intervention.
  The Verbal Fluency Task is a neuropsychological measure of lexical retrieval efficiency and executive functioning. In this test, the participants are asked to name the words that starts with a specific alphabet (phonemic fluency) in 60 seconds. The verbal fluency score is calculated based on the number of correct/acceptable words produced within the allotted time.

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Parikh, PhD, Principal Investigator — Temple University; Jason Chein, PhD, Principal Investigator — Temple University; Tania Giovannetti, PhD, Principal Investigator — Temple University
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No